CLINICAL TRIAL: NCT02240602
Title: Optimal Dose of i.v Oxycodone for Postoperative Pain After Laparoscopic Colorectal Surgery
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Lack of internal resources
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OxyNorm
Record Dates: First submitted 2014-09-11; First posted 2014-09-15 (Estimated); Last update posted 2015-06-16 (Estimated); Status verified 2014-09

CONDITIONS: Pain
Keywords: acute pain; postoperative; surgery
MeSH Terms: conditions — Pain; Acute Pain | interventions — Oxycodone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Oxycodone, 1.00 mg dose (Experimental): Regimen of intravenous patient-controlled analgesia consists of bolus dose of oxycodone 1.00 mg with lock out time of 10 min without basal infusion.
  Interventions: Drug: Oxycodone, 1.00 mg dose
- Oxycodone, 0.03 mg/kg dose (Experimental): Regimen of intravenous patient-controlled analgesia consists of bolus dose of oxycodone 0.03 mg/kg with lock out time of 10 min without basal infusion.
  Interventions: Drug: Oxycodone, 0.03 mg/kg dose
- Oxycodone, 0.02 mg/kg dose (Experimental): Regimen of intravenous patient-controlled analgesia consists of bolus dose of oxycodone 0.02 mg/kg with lock out time of 10 min without basal infusion.
  Interventions: Drug: Oxycodone, 0.02 mg/kg dose

INTERVENTIONS:
Drug: Oxycodone, 1.00 mg dose — Intravenous oxycodone is provided as patient-controlled analgesia after surgery with bolus dose of 1.00 mg.
  Other Names: OxyNorm
  Arms: Oxycodone, 1.00 mg dose
Drug: Oxycodone, 0.03 mg/kg dose — Intravenous oxycodone is provided as patient-controlled analgesia after surgery with bolus dose of 0.03 mg/kg.
  Other Names: OxyNorm
  Arms: Oxycodone, 0.03 mg/kg dose
Drug: Oxycodone, 0.02 mg/kg dose — intravenous oxycodone is provided as patient-controlled analgesia after surgery with bolus dose of 0.02 mg/kg.
  Other Names: OxyNorm
  Arms: Oxycodone, 0.02 mg/kg dose

SUMMARY:
Postoperative pain control is required after major abdominal surgery, including laparoscopic colorectal surgery. Intravenous oxycodone is widely used for postoperative acute pain control mainly in Europe. The aim of this study is to evaluate the optimal dose of intravenous oxycodone for pain control after laparoscopic colorectal surgery in Korean.

DETAILED DESCRIPTION:
Oxycodone is known to be effective in pain control and has less sedative effect than morphine does. It has been described that distribution of cytochrome P450, which is associated with metabolism of oxycodone, differed between the races. Proper dose of intravenous oxycodone after major abdominal surgery has not been well defined in Korean. The purpose of this study is to evaluate the optimal dose of intravenous oxycodone for pain control after laparoscopic colorectal surgery in Korean based on pain score and side effects.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists class 1,2
* Expected surgical time between 2 - 6 hours
* Scheduled for laparoscopic colorectal surgery

Exclusion Criteria:

* Severe dysfunction of liver, heart, kidney, or lung
* Cannot understand numeric rating scale of pain
* Known or suspected allergy to oxycodone
* Previous history of postoperative nausea or vomiting
* Medication of antidepressants
* Postoperative long-term ICU care or prolonged mechanical ventilatory support
* Chronic pain
* Drug abuser
* Hypersensitivity reaction to aspirin or NSAIDs
* Refuse to enroll

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-07; Primary Completion 2016-10 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
resting postoperative pain at 24hr | 24 hr after surgery
  Primary outcome is resting postoperative pain at 24 hr after surgery with numeric rating scale 0-10.

SECONDARY OUTCOMES:
side effects | 24 hr after surgery
  Secondary outcome includes any side effect at 24 hr after surgery.

OTHER OUTCOMES:
sedation | 24 hr after surgery
  sedation with Ramsay sedation score (1-6) at 24 hr after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Yunseok Jeon, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea